CLINICAL TRIAL: NCT03619850
Title: A Phase 3, Randomized, Open-Label, Multicenter Study to Evaluate the Safety (Compared to Iron Sucrose), Efficacy and Pharmacokinetics of Ferumoxytol for the Treatment of Iron Deficiency Anemia (IDA) in Pediatric Subjects With Chronic Kidney Disease (CKD)
Brief Title: A Study to Evaluate the Safety (Compared to Iron Sucrose), Efficacy and Pharmacokinetics of Ferumoxytol for the Treatment of Iron Deficiency Anemia (IDA) in Pediatric Subjects With Chronic Kidney Disease (CKD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-FER-CKD-354
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease; Iron Deficiency Anemia
Keywords: Iron deficiency anemia (IDA); chronic kidney disease (CKD); pediatrics; ferumoxytol; iron sucrose; Feraheme; Venofer
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferumoxytol (Experimental)
  Interventions: Drug: Ferumoxytol
- Iron sucrose (Active Comparator)
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Ferumoxytol — Each 20 mL single-use vial contains 17 mL of ferumoxytol that consists of iron at a concentration of 30 mg Fe/mL, coated with polyglucose sorbitol carboxymethylether and formulated with mannitol, at a concentration of 44 mg/mL, in a black to reddish brown sterile, aqueous, colloidal, isotonic solution.
  Other Names: Feraheme
  Arms: Ferumoxytol
Drug: Iron sucrose — Each mL contains 20 mg of elemental iron as iron sucrose in water for injection. The 5 mL single-use vial contains 100 mg of iron per 5 mL. The drug product contains approximately 30% sucrose (300 mg/mL).
  Other Names: Venofer
  Arms: Iron sucrose

SUMMARY:
Primary Objectives:

To evaluate the safety (compared to iron sucrose) and efficacy of ferumoxytol in pediatric CKD subjects with iron deficiency anemia (IDA) or who are at risk of development of IDA

Secondary Objective:

To determine the single-dose pharmacokinetics (PK) and pharmacodynamics (PD) profile of ferumoxytol in pediatric subjects.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, open-label, multicenter, study of the safety (compared to iron sucrose), efficacy, and PK/PD of ferumoxytol (7.0 mg Fe/kg x 2 [max 510 mg/dose]) in pediatric subjects with iron deficiency anemia (IDA) and CKD. There will be a total of approximately 125 subjects randomized to treatment in a 2:1 ratio to either ferumoxytol or iron sucrose.

Total subject participation in the study will be up to 7 weeks, which includes a 2-week Screening Period and a 5-week Treatment Period.

Subjects receive the following:

• Two IV infusions of ferumoxytol 7.0 mg Fe/kg (max 510 mg/dose), the first administered on Day 1 and the second 2-8 days later

OR

• Iron sucrose (Venofer®): For Hemodialysis Dependent (HDD) patients: 2 mg Fe/kg, administered on consecutive dialysis sessions, for 10 doses (max 100mg/dose with a total max treatment course of 1000mg) For Non-hemodialysis Dependent (NDD) or Peritoneal Dialysis De pendent(PDD) patients: 4 mg Fe/kg, administered up to 3 times/week, for 5 doses (max 200mg/dose with a total max treatment course of 1000mg).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 2 years to <18 years of age at time of consent
2. Has IDA defined as: a) hemoglobin <12.0 g/dL and b) with either transferrin saturation (TSAT) <40% or ferritin <100 ng/mL; or considered to be at risk of development of IDA, i.e., TSAT<20% with falling hemoglobin during the preceding 2 months and a history of hemoglobin <12 g/dL
3. Has Chronic Kidney Disease defined as one of the following:

   1. on chronic hemodialysis;
   2. receiving chronic peritoneal dialysis;
   3. estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73 m2;
   4. has evidence of structural and/or functional abnormalities e.g., persistent albuminuria, abnormal urine sediment, electrolyte and other abnormalities due to tubular disorders for > 3 months.
4. For patients other than hemodialysis dependent CKD patients, documented history of unsatisfactory oral iron therapy or in whom oral iron cannot be tolerated, or for whom oral iron is considered medically inappropriate
5. All subjects (female and male) of childbearing potential who are sexually active must be on an effective method of birth control for at least 1 month prior to Day 1 Dosing and agree to remain on birth control until completion of the study

Exclusion Criteria:

1. Known hypersensitivity reaction to any component of ferumoxytol and iron sucrose
2. History of allergy to intravenous (IV) iron
3. History of multiple drug allergies (>2)
4. Low systolic blood pressure (Age 1-9 years <70 + [age in years x 2] mmHg, Age 10-17 years <90 mmHg)
5. Hemoglobin ≤7.0 g/dL
6. Serum ferritin level >600 ng/mL

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin change of at least 0.5 g/dL from Baseline to Week 5 | 35 days
  Proportion of patients achieving a hemoglobin change of at least 0.5 g/dL during the period from Baseline to Week 5

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | 49 days
  Incidence of Treatment Emergent Adverse Events
Incidence of adverse events of special interest (AESI) | 49 days
  Incidence of adverse events of special interest (AESI) (hypotension and hypersensitivity)

OTHER OUTCOMES:
Area Under the Curve (AUC) | 35 days
  Pharmacokinetic parameter: Area Under the Curve (AUC)
Clearance | 35 days
  Pharmacokinetic parameter: clearance
Distribution and elimination half-lives | 35 days
  Pharmacokinetic parameter: distribution and elimination half-lives

CONTACTS AND LOCATIONS:
Locations (21):
- United States (8):
  - Memorial Healthcare System, Hollywood, Florida
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - The Feinstein Institute Medical Research Organization of Northwell Health, Inc., Lake Success, New York
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Mount Sinai Hospital (MSH), New York, New York
  - Montefiore Medical Center (MMC) - The Children's Hospital at Montefiore (CHAM), The Bronx, New York
  - Akron Nephrology Associates, Inc., Akron, Ohio
  - West Virginia University, Morgantown, West Virginia
- Hungary (2):
  - Semmelweis Egyetem - Altalanos Orvostudomanyi Kar (SE AOK) - I. sz. Gyermekgyogyaszati Klinika, Budapest
  - University Of Szeged, Szeged
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Klaipeda Children's Hospital, Klaipėda
  - Vsl Vilniaus Universiteto Vaiku Ligonine (VUVL) (Vilnius University Children's Hospital), Vilnius
- Mexico (4):
  - Instituto Mexicano De Trasplantes S.C, Cuernavaca
  - JM Research, SC, Cuernavaca
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Instituto Nacional de Pediatria (INP) (National Institute of Pediatrics), Mexico City
- Poland (4):
  - Uniwersytecki Szpital Kliniczny Im. Zamenhofa w Bialystoku, Bialystok
  - Specjalistyczne Gabinety Sp. z o.o, Krakow
  - University Children Hospital, Krakow
  - Polish Mother's Memorial Hospital Research Institute, Lodz

IPD SHARING:
Plan to Share IPD: No